CLINICAL TRIAL: NCT00060385
Title: Diffuse Large B Cell And Peripheral T Cell Non-Hodgkin's Lymphomas (NHL) In The Elderly. Influence Of Prolonged Oral Etoposide Added To CHOP Combination Chemotherapy In Patients With Good Physiological Status. An EORTC Randomized Phase II-III Trial Including Geriatric Assessment And Quality Of Life
Brief Title: Combination Chemotherapy With or Without Etoposide in Treating Older Patients With Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-20991; EORTC-20991
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lymphoma
Keywords: stage I adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II adult T-cell leukemia/lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Large B-Cell, Diffuse | interventions — VAP-cyclo protocol; EPOCH protocol; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: CHOP regimen
Drug: EPOCH regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating non-Hodgkin's lymphoma.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of combination chemotherapy with or without etoposide in treating older patients who have non-Hodgkin's lymphoma that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the complete response rates in older patients with diffuse large B-cell or peripheral T-cell non-Hodgkin's lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) with vs without etoposide.
* Compare the overall survival of patients treated with these regimens.
* Compare the time to treatment failure in patients treated with these regimens.
* Compare the freedom from progression in patients treated with these regimens.
* Determine the toxicity of CHOP plus etoposide in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to cellular type (B-cell vs T-cell), initial stage of disease (I and II vs III and IV), WHO performance status (0-1 vs 2), and lactic dehydrogenase level (LDH) (normal vs abnormal). Patients are randomized to 1 of 2 treatment arms.

* Arm I (CHOP chemotherapy): Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1. Patients also receive oral prednisone on days 1-5. Treatment repeats every 21 days for 3 courses in the absence of unacceptable toxicity. Patients then undergo disease evaluation.

Patients with disease progression or no change in disease are removed from study. Patients with responsive stage I or II disease receive 1 additional course if they demonstrate all 3 of the following conditions (at baseline): no LDH elevation, WHO performance status of 0-1, and greatest single diameter of any tumor site less than 5 cm. Patients with responsive stage I or II disease receive 3 additional courses if they demonstrate 1 or more of the following conditions (at baseline): LDH elevation, WHO performance status 2, and/or greatest single diameter of any tumor site at least 5 cm. Patients with responsive stage III or IV disease receive 3 additional courses.

After the completion of chemotherapy, patients with responsive stage I or II disease undergo involved field radiotherapy once daily 5 days a week for 3.5-4 weeks. Patients with initial bulky stage III or IV disease may also undergo radiotherapy.

* Arm II (CHOP chemotherapy and etoposide): Patients receive CHOP chemotherapy as in arm I plus oral etoposide 2 or 3 times daily on days 1-10. Treatment repeats every 21 days for 3 courses in the absence of unacceptable toxicity. Patients receive additional courses as in arm I.

After the completion of chemotherapy, patients with responsive stage I or II disease or initial bulky stage III or IV disease undergo radiotherapy as in arm I.

Quality of life is assessed at baseline, after course 3, at the end of chemotherapy, every 6 months for 3 years, and then annually thereafter.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 686 patients (126 for phase II and 560 for phase III) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell* or peripheral T-cell non-Hodgkin's lymphoma by REAL/WHO classification, including the following:

  * All morphological and clinical variants
  * All Ann Arbor stages NOTE: *Presence of a small cell, indolent lymphoma component in the bone marrow biopsy is allowed
* No Burkitt-like lymphoma
* Previously untreated disease
* No cerebral or meningeal involvement
* At least 1 measurable target lesion at least 1.1 cm by the Cheson criteria

PATIENT CHARACTERISTICS:

Age

* 70 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3 (unless related to bone marrow infiltration)

Hepatic

* Bilirubin less than 1.8 mg/dL*
* AST or ALT less than 2.5 times upper limit of normal (ULN)*
* Alkaline phosphatase less than 4 times ULN* NOTE: *Values above these thresholds are allowed only if related to non-Hodgkin's lymphoma

Renal

* Creatinine clearance at least 50 mL/min

Cardiovascular

* LVEF at least 50%

Other

* HIV negative
* No history of concurrent severe disease that would preclude study treatment
* No other prior or concurrent malignancy except adequately treated basal cell skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid malignancy with no evidence of disease for at least 5 years prior to study entry
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent participation in another investigational drug study
* No other concurrent antineoplastic agents

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-03; Primary Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Soubeyran, MD, PhD, Study Chair — Institut Bergonié
Locations (1):
- U.Z. Gasthuisberg, Leuven, Belgium